CLINICAL TRIAL: NCT02101840
Title: Abuse Liability of Controlled-Release Oxycodone Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Beth Sproule, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 043-2013
Record Dates: First submitted 2014-03-24; First posted 2014-04-02 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Substance-Related Disorders
Keywords: Substance-Related Disorders; Prescription Drug Misuse; Analgesics, Opioid; Oxycodone; Randomized Controlled Trial; Cross-Over Studies; Placebo; Healthy Volunteers
MeSH Terms: conditions — Substance-Related Disorders; Prescription Drug Misuse | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apo-Oxycodone CR® (Active Comparator): a single 40mg oral dose of the controlled release oxycodone formulation Apo-Oxycodone CR®
  Interventions: Drug: Apo-Oxycodone CR®
- OxyNEO® (Active Comparator): a single 40mg oral dose of the controlled release oxycodone formulation OxyNEO®
  Interventions: Drug: OxyNEO®
- Placebo (Placebo Comparator): a single oral dose of placebo prepared using gelatin capsules and lactose filler with identical looking study capsules as the oxycodone products
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apo-Oxycodone CR® — a single 40mg oral dose of the controlled release oxycodone formulation Apo-Oxycodone CR®
  Other Names: Oxycodone
  Arms: Apo-Oxycodone CR®
Drug: OxyNEO® — a single 40mg oral dose of the controlled release oxycodone formulation OxyNEO®
  Other Names: Oxycodone
  Arms: OxyNEO®
Drug: Placebo — a single oral dose of placebo prepared using gelatin capsules and lactose filler with identical looking study capsules as the oxycodone products
  Arms: Placebo

SUMMARY:
The objective of this study is to examine the abuse liability of a single 40mg dose of 2 controlled release oxycodone formulations (Apo-Oxycodone CR® and OxyNEO®) in non-dependent recreational opioid users by assessing the self-reported acute effects of the drugs and taking blood samples to measure drug concentrations. The investigators think there may be differences in how well these drugs are liked when swallowed whole due to differences in how the products are formulated.

DETAILED DESCRIPTION:
This is a single-center, single-dose, double-blind, placebo-controlled, randomized, crossover, abuse liability study conducted in healthy subjects who are non-dependent recreational opioid users. The study consists of 3 study days during which each subject will take one tablet of either 40mg OxyNEO®, 40mg Apo-Oxycodone CR®, or placebo. The participants will be assessed for both pharmacokinetic and pharmacodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to 50 years of age
* Willing and capable to give written informed consent
* Subjects must have used opioids recreationally to achieve a "high" on at least five occasions in the 12 months before screening and at least once in the 90 days before screening according to self-report
* Females of childbearing potential have to use a medically acceptable form of birth control and have a negative pregnancy test
* Pass medical assessment, which includes physical examination, assessment of medical history, vital signs, blood work, and urine toxicology screen
* Willing to abstain from alcohol 12 hours before and during the study days

Exclusion Criteria:

* Current or past Axis I psychiatric illness (including current drug dependence or past opioid dependence, except nicotine dependence)
* Current hepatic disease or renal failure
* Pregnancy or lactation in women
* Current medication that is known to interact with opioids
* Known contraindications or hypersensitivity to opioids
* Current opioid therapy
* Chronic pain disorder requiring regular medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Visual Analogue Scale for "Drug Liking" Over 8 Hours After Drug Administration | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Change from Baseline on Visual Analogue Scale for "Drug High" Over 8 Hours After Drug Administration | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration

SECONDARY OUTCOMES:
Pupil Diameter | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Cmax | Baseline to 6 hours post-administration
  Plasma oxycodone concentration
Profile of Mood States (POMS) | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Psychomotor Performance | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Digit Symbol Substitution Test (DSST)
Visual Analogue Scale for "Any Drug Effects" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Good Effects" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Bad Effects" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Feel Sick" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Nausea" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Sleepy" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Visual Analogue Scale for "Dizzy" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Sedation | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Euphoria | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Dysphoric Changes | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Psychotomimetic Changes | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Somatic Disturbances | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Sensory Disturbances | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
  Addiction Research Center Inventory (ARCI)
Tmax | Baseline to 6 hours post drug administration
  Plasma oxycodone concentrations
Visual Analogue Scale for "Take Drug Again" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration
Likert Scale for "Sedation" | Baseline and 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Beth Sproule, PharmD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research